CLINICAL TRIAL: NCT01110642
Title: Open-label, Pilot Study to Assess Cholesterol-Lovastatin Solution in the Treatment of Syndromic Ichthyoses
Brief Title: Novel Treatment for Syndromic Ichthyoses
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was withdrawn due to lack of eligible population for study
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Professor and Chair of Department of Dermatology, Professor of Pediatrics, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-04-15
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Syndromic Ichthyoses; CHILD Syndrome; Smith Lemli Opitz Syndrome; Conradi Syndrome
MeSH Terms: conditions — Congenital Hemidysplasia with Ichthyosiform Erythroderma and Limb Defects; Smith-Lemli-Opitz Syndrome | interventions — Lovastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lovastatin solution (Experimental): All patients will receive lovastatin solution
  Interventions: Drug: Lovastatin

INTERVENTIONS:
Drug: Lovastatin — Topical lovastatin applied to red, rashy areas two times daily for 12 months

SUMMARY:
This is an open label-pilot study to assess the efficacy and safety of a novel cholesterol-lovastatin topical solution in children with rare syndromic ichthyoses. Often times, these children have difficulty in finding easily applied treatments to make their psoriasiform and ichthyotic plaques more manageable. We propose the use of a cholesterol-lovastatin topical solution as a treatment option with the hypothesis that it will lead to regression of involved areas and decreased erythema and warty-like appearance of the plaques. We plan to enroll children with syndromic ichthyoses over the age of 1 year for a 12 month study with a total of 5 visits and 5 phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent form signed by the subject or subject's legal representative; also, if the subject is under the age of majority but capable of providing assent, signed assent from the subject.
* Diagnosis of a syndromic ichthyoses (verified by Dr Amy S. Paller).
* Children and adults 12 months of age and above

Exclusion Criteria:

* Use of any investigational drug within the 30 days before enrollment.
* Current malignancy.
* Pregnancy or breastfeeding during the study. (All female subjects of childbearing potential will be assessed for pregnancy at all visits.)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07

PRIMARY OUTCOMES:
Physician global assessment of severity (PGAS) | 12 months
  Difference in physician global assessment of severity at baseline compared to month 12

SECONDARY OUTCOMES:
Total body surface area (TBSA) | 12 months
  Percent change in TBSA affected at baseline compared to at month 12

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Paller, MD, Principal Investigator — Northwestern University